CLINICAL TRIAL: NCT04432766
Title: A Phase 1/2, Multi-Center, Randomized Study to Assess Safety, Pharmacokinetics, Immunogenicity, and Efficacy of BAT2020 in Hospitalized Patients Infected With SARS-CoV-2 (COVID-19)
Brief Title: A Phase 1/2 Study to Assess Safety and Efficacy of BAT2020 in Hospitalized COVID-19 Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: strategic decision
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAT-2020-001-CR
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose (Experimental)
  Interventions: Drug: BAT2020
- Medium dose (Experimental)
  Interventions: Drug: BAT2020
- High dose (Experimental)
  Interventions: Drug: BAT2020

INTERVENTIONS:
Drug: BAT2020 — After a cohort completes the study on Day 28, data on safety and tolerability for each cohort will be evaluated by the Safety Monitoring Committee (SMC). Administration of the next higher dose to a new dosing cohort will be permitted only if adequate safety and tolerability have been demonstrated. If encouraging clinical benefit is observed at a certain dose level, the study may proceed to a to Part 2 based on emerging data.

SUMMARY:
This is a randomized study to assess safety, pharmacokinetics, immunogenicity, and efficacy of BAT2020 in hospitalized patients infected with COVID-19. This study is composed of 2 Parts: a single ascending dose (Part 1) and single dose(s) tested in parallel with a double-blind, placebo-controlled design (Part 2). Patients also will receive best available standard of care (SOC) treatment. A data and safety monitoring board (DSMB) will be set up for the study.

ELIGIBILITY:
1. Male or nonpregnant female adult ≥18 years of age at time of enrollment.
2. Patient (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
3. Agrees to the collection of nasopharyngeal swabs for virology assessment.
4. Women of childbearing potential must agree to either abstinence or use at least 1 primary form of contraception at the time of screening and for 4 months after study drug dosing.
5. Enrollment within 72 hours of hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-20 (Estimated); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-08-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Day 28
  SAE, TEAEs, mortality, those resulting in treatment discontinuation, and changes from baseline in safety laboratory assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Snake River Research, Idaho Falls, Idaho, United States